CLINICAL TRIAL: NCT01496391
Title: A Single Centre Open Label Comparison of [I-123]-Ortho-Iodohippuric Acid (OIH) With [Tc-99m]-Mercaptoacetyltriglycine (MAG3) for Assessment of Renal Tubular Function
Status: Completed | Type: Observational
Sponsor: Centre for Probe Development and Commercialization (Other)
Collaborators: McMaster University (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Other Study IDs: CPDC-HIPP-001
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Renal Function Impairment
Keywords: imaging; renal function; I-123 OIH; Tc-99m MAG 3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood (chemistry, hematology) and kidney function (eGRF, eRPF)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy Participants: eGFR ≥60 ml/min/1.73m^2, healthy prospective kidney donor
- Moderate Renal Function Impairment: eGFR 30-59 ml/minute/1.73m^2
- Severe Renal Function Impairment: eGFR <30 mL/minute/1.73m^2

SUMMARY:
Iodine-123 labelled ortho-Iodohippuric Acid ([I-123]-OIH) was used in the early 1970's as a kidney imaging agent or tracer that "lights-up" inside your body when scanned, but over the years its use has declined. The most commonly used tracer is Technetium-99m labelled Mercaptoacetyltriglycine ([Tc-99m]-Mertiatide or [Tc-99m]-MAG3). However, long-term shortages may threaten the supply of the radioactive substance Tc-99m in Canada and the world. As a result of such shortages, there is a need to identify other types of tracers that can be used for imaging. [I-123]-OIH may be an alternative.

The purpose of this study is to examine the diagnostic performance characteristics of [I-123]-OIH in comparison to [Tc-99m]-MAG3.

DETAILED DESCRIPTION:
This study is being conducted to compare two imaging agents (tracers): [I-123]-OIH and [Tc-99m]-MAG3 using gamma camera imaging in participants with different levels of kidney function. Gamma camera imaging is a non-invasive nuclear scan that is used to look at organs and tissues inside the body. An imaging agent or tracer is a radioactive chemical intravenously injected into your body which lights up cells, tissues and organs. The study will evaluate the safety of a single injection of [I-123]-OIH and compare the imaging results and the calculated renal function values (using blood tests) to those of [Tc-99m]-MAG3 . 90 participants are required to complete this study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Provide signed informed consent.
* Documented stable renal impairment with an eGFR < 60/mL/min/1.73m^2 by two eGFR measurements within 3 months that are within ± 15% of each other or healthy prospective kidney donor with an eGFR ≥ 60 mL/min/1.73m^2.

Exclusion Criteria:

* Females who are pregnant, planning to become pregnant or are lactating.
* Clinically relevant abnormal findings that could, in the opinion of the investigator, interfere with the safe completion of the study.
* Unable, in the opinion of the clinician or investigator, to tolerate fluid intake required for radionuclide renography.
* Participation in any clinical trial involving an investigational product within 30 days prior to the first injection.
* Not using an adequate method of family planning unless the participant, or the male participant's partner, has had a hysterectomy, a tubal ligation, is postmenopausal or is not at risk of pregnancy.
* Unable to lie still in a supine position for at least 30 minutes.
* Unable to complete study procedures, including follow-up safety assessments.
* Medical or psychological conditions that on assessment by the principal investigator make the participant unable to complete the procedure.
* History of allergic reaction to iodine or iodine compounds, inclusive of iodinated x-ray contrast media.
* Any other conditions that may impact the participant's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from both healthy subjects (eGFR ≥ 60 mL/minute/1.73m^2) being assessed as potential renal donors and patients having suspected renal impairment (eGFR <60 mL/minute/1.73m^2). Severity of disease will be determined based on estimated glomerular filtration rate (eGFR) derived from serum creatinine concentration.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
[I-123]-OIH Safety | Visit 3 and Follow-up Phone Call
  Evaluate the safety of a single injection of [I-123]-OIH administered to a population of healthy prospective kidney donors and patients with stable chronic renal impairment.
Compare kidney function using [I-123]-OIH and [Tc-99m]-MAG3 imaging | Visit 2 and 3
  Compare results of renal plasma flow derived from [I-123]-OIH and [Tc-99m]-MAG3 gamma camera images of healthy prospective kidney donors and patients with stable chronic renal impairment.

SECONDARY OUTCOMES:
Qualitative Assessment | Visit 2 and 3
  Compare the qualitative assessment of kidney uptake, urine excretion and image quality of [I-123]-OIH and [Tc-99m]-MAG3 in an independent read by two nuclear medicine physicians blinded to all participant clinical data.
Image-derived Perfusion Data | Visits 2 and 3
  Compare results of differential perfusion(from image-derived perfusion data) of [I-123]-OIH and [Tc-99m]-MAG3.
eRPF | Visits 2 and 3
  Compare results of effective renal plasma flow (eRPF), using the single sample clearance method of [I-123]-OIH and [Tc-99m]-MAG3.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gulenchyn, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joesph's Healthcare Hamilton, Hamilton, Ontario, Canada